CLINICAL TRIAL: NCT04388826
Title: Randomized, Placebo-Controlled, Phase 2 Study of VERU-111 for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) in Patients at High Risk for Acute Respiratory Distress Syndrome (ARDS)
Brief Title: COVID-19 Treatment of Severe Acute Respiratory Syndrome With Veru-111
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veru Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V0211901
Record Dates: First submitted 2020-05-13; First posted 2020-05-14 (Actual); Results first posted 2021-11-24 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — sabizabulin

STUDY DESIGN:
Intervention Model Description: Randomized Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind Randomized Placebo-Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Veru-111 18 mg (Experimental): Veru-111 18mg capsules
  Interventions: Drug: Veru-111
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Drug: Veru-111

INTERVENTIONS:
Drug: Veru-111 — Respiratory Distress Syndrome, Adult
  Other Names: Bisindole

SUMMARY:
To demonstrate the efficacy of VERU-111 in the treatment of SARS-Cov-2 Infection by assessing its effect on the proportion of subjects that are alive without respiratory failure at Day 22. Respiratory failure is defined as non-invasive ventilation or high-flow oxygen, intubation and mechanical ventilation, or ventilation with additional organ support (e.g., pressors, RRT, ECMO).

DETAILED DESCRIPTION:
This study is a multicenter, randomized, placebo-control, efficacy and safety study of VERU-111 for the treatment of COVID-19. Subjects will receive either 18 mg of VERU-111 or matching placebo orally or through nasogastric tube daily for to 21 days or until the subject is discharged from the hospital, whichever comes first.

The primary efficacy endpoint of the study will be the proportion of subjects that are alive without respiratory failure at Day 22. Respiratory failure is defined as non-invasive ventilation or high-flow oxygen, intubation and mechanical ventilation, or ventilation with additional organ support (e.g., pressors, RRT, ECMO).

The total study duration for a subject from screening to follow up visit is planned to be 62 days.

An evaluation of the effect of VERU-111 on SARS-CoV-2 (COVID-19) compared to the placebo control will be evaluated after the last subject has completed Day 22. This will allow for the decision to move to Phase 3 more quickly if the Phase 2 portion of the study shows a clinically relevant difference in the proportion of subjects that are alive without respiratory failure at Day 22 in the VERU-111 treated groups compared to the Placebo treatment group and VERU-111 is well tolerated in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent
2. Be able to communicate effectively with the study personnel
3. Aged ≥18 years
4. Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) infection confirmed by polymerase chain reaction (PCR) test
5. Patients at high risk for ARDS, with known comorbidities for being at high risk, such as, Asthma (moderate to severe), Chronic Lung Disease, Diabetes, Chronic Kidney Disease being treated with dialysis, Severe Obesity (BMI ≥40), 65 years of age or older, primarily reside in a nursing home or long-term care facility, immunocompromised
6. Peripheral capillary oxygen saturation (SpO2) ≤ 94% on room air at screening
7. Subjects must agree to use acceptable methods of contraception

   * If subject is female or the male subject's partner could become pregnant, use acceptable methods of contraception from the time of the first administration of study medication until 6 months following administration of the last dose of study medication. Acceptable methods of contraception are as follows: Condom with spermicidal foam/gel/film/cream/suppository [i.e., barrier method of contraception], surgical sterilization (vasectomy with documentation of azospermia) and a barrier method {condom used with spermicidal foam/gel/film/cream/suppository}, the female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or subdermal implants and a barrier method (condom used with spermicidal foam/gel/film/cream/suppository)
   * If female subject or the female partner of a male subject has undergone documented tubal ligation (female sterilization), a barrier method (condom used with spermicidal foam/gel/film/cream/suppository) should also be used
   * If female subject or the female partner of a male subject has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS), a barrier method (condom with spermicidal foam/gel/film/cream/suppository) should also be used
8. Subject is willing to comply with the requirements of the protocol through the end of the study

Exclusion Criteria:

1. Known hypersensitivity or allergy to colchicine
2. Participation in any other clinical trial of an experimental treatment for COVID-19
3. Concurrent treatment with other experimental agents with actual or possible direct acting antiviral activity against COVID-19 is prohibited < 24 hours prior to study drug dosing (except standard of care) Remdesivir and convalescent plasma is allowed as standard of care.
4. Requiring mechanical ventilation at screening
5. Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) >2 X upper limit of normal (ULN)
6. Total bilirubin > ULN
7. Creatinine clearance < 60 mL/min
8. Documented medical history of liver disease, including but not limited to, prior diagnosis of hepatitis of any etiology, cirrhosis, portal hypertension, or confirmed or suspected esophageal varices
9. Moderate to severe renal impairment
10. Hepatic impairment
11. Positive for HbsAg, or HCV antibodies at screening
12. Any comorbid disease or condition (medical or surgical) which might compromise the hematologic, cardiovascular, endocrine, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk
13. Participants must agree to refrain from prolonged exposure to the sun or agree to use at least SPF 50 on all exposed skin and protective clothing during prolonged sun exposure throughout participation in this study and/or treatment with VERU-111.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barnette, Study Director — Veru Inc.
Locations (5):
- United States (5):
  - HonorHealth, Scottsdale, Arizona
  - Methodist Hospital, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Inspira Medical Center, Vineland, New Jersey
  - Memorial Hermann Memorial City Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Veru-111 18 mg QD: Veru-111 18mg capsules
  Veru-111: Respiratory Distress Syndrome, Adult
- Placebo QD: Placebo capsules
  Veru-111: Respiratory Distress Syndrome, Adult
Period: Overall Study
Arm/Group | Veru-111 18 mg QD | Placebo QD
Started | 19 | 20
Completed | 15 | 18
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Number of Patients Exposed to Veru-111 18 mg: Veru-111 18mg capsules
  Veru-111: Respiratory Distress Syndrome, Adult
- Number of Patients Exposed to Placebo: Placebo capsules
  Veru-111: Respiratory Distress Syndrome, Adult
- Total: Total of all reporting groups
Arm/Group | Number of Patients Exposed to Veru-111 18 mg | Number of Patients Exposed to Placebo | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (11.40) | 57.8 (13.32) | 58.5 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 10 | 17 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 19 | 16 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Are Alive Without Respiratory Failure at Day 29.
Description: To demonstrate the efficacy of VERU-111 in the treatment of SARS-Cov-2 Infection by assessing its effect on the proportion of subjects that are alive without respiratory failure at Day 29. Respiratory failure is defined as endotracheal intubation and mechanical ventilation, extracorporeal membrane oxygenation, high-flow nasal cannula oxygen delivery, noninvasive positive pressure ventilation, clinical diagnosis of respiratory failure with initiation of none of these measures only when clinical decision making is driven solely by resource limitation
Time Frame: Day 29
Population: Responders
Measure: Count of Participants; unit: Participants
Arm/Group | Veru-111 18 mg | Placebo
Number analyzed (Participants) | 19 | 20
Participants | 17 | 14

2. Secondary Outcome: World Health Organization Ordinal Scale Clinical Improvement
Description: Improvement on the World Health Organization Ordinal Scale for Clinical Improvement. 8-point ordinal scale (WHO scale from 0 to 8). Lower value equals better while higher value equals worse
  Score of 0 Uninfected No clinical or virologic evidence of infection Score of 1 Ambulatory No limitation of activities Score of 2 Limitation of activities Score of 3 Hospitalized, no oxygen therapy Score of 4 Oxygen by mask or nasal prongs Score of 5 Non-invasive ventilation or high-flow oxygen Score of 6 Intubation and mechanical ventilation Score of 7 Ventilation + additional organ support - pressors, RRT, ECMO Score of 8 Death
Time Frame: Day 29
Population: World Health Organization Ordinal Scale for clinical improvement (Eight Point Ordinal Scale)-With Last Observation Carried Forward Values
Measure: Mean (Standard Deviation); unit: Units on WHO COVID Scale
Arm/Group | Veru-111 18 mg | Placebo
Number analyzed (Participants) | 19 | 20
Units on WHO COVID Scale | -1.7 (1.49) | -1.1 (2.42)

3. Secondary Outcome: Proportion of Subjects With Fever Normalization and SPO2 Greater Than 94% by Visit
Description: Proportion of subjects with normalization of fever and oxygen saturation through. Responders are subjects who have been discharged from the hospital or has fever normalization maintained for at least 24 hours AND peripheral capillary oxygen saturation (SPO2) greater than 94% sustained for 24 hours is observed at the time of the visit.
  Non-responders are subjects who died before the visit or do not meet both criteria of the end point at the time of the visit.
Time Frame: Day 15, Day 22 and Day 29
Population: Responders are subjects who have been discharged from the hospital or has fever normalization maintained for at least 24 hours AND peripheral capillary oxygen saturation (SPO2) greater than 94% sustained for 24 hours is observed at the time of the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Veru-111 18 mg QD | Placebo QD
Number analyzed (Participants) | 19 | 20
Participants
  Day 15 | 14 | 12
  Day 22 | 17 | 16
  Day 29 | 17 | 14

4. Secondary Outcome: Proportion of Subjects Alive and Discharged From Hospital by Visit
Description: Proportion of subjects alive and discharged from hospital by visit. Responders are subjects who are alive and have been discharged from the hospital at the time of the visit. (Non-responders are subjects who died before the visit or in the hospital at the time of the visit).
Time Frame: Day 15, Day 22 and Day 29
Population: Responders - subjects who are alive and have been discharged from the hospital at the time of the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Veru-111 18 mg QD | Placebo QD
Number analyzed (Participants) | 19 | 20
Participants
  Day 15 | 14 | 12
  Day 22 | 17 | 15
  Day 29 | 18 | 14

5. Secondary Outcome: Patients Alive and Free of Respiratory Failure
Description: Proportion of patients alive and free or respiratory failure
Time Frame: Day 15 and Day 22
Population: Responders
Measure: Count of Participants; unit: Participants
Arm/Group | Veru-111 18 mg QD | Placebo QD
Number analyzed (Participants) | 19 | 20
Participants
  Day 15 | 16 | 13
  Day 22 | 16 | 14

ADVERSE EVENTS:
Time Frame: 62 Days
Arm/Group | Veru-111 18 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/19 | 5/20
Serious Adverse Events (participants affected / at risk) | 3/19 | 5/20
Other Adverse Events (participants affected / at risk) | 12/19 | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veru-111 18 mg (N=19) | Placebo (N=20)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Septic Sock (Infections and infestations) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veru-111 18 mg (N=19) | Placebo (N=20)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2)
Septic Shock (Infections and infestations) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT04388826/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT04388826/SAP_002.pdf